CLINICAL TRIAL: NCT00842946
Title: Exposure With Acceptance-Based Versus Habituation-Based Rationale for Public Speaking Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Responsible Party: Principal Investigator, James Herbert, Professor of Psychology, Drexel University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DRX-17819
Record Dates: First submitted 2009-02-11; First posted 2009-02-12 (Estimated); Results first posted 2014-06-02 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: Public Speaking; Social Fear
MeSH Terms: conditions — Speech

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exposure w/ Acceptance-Based Rationale (Experimental): Behavioral exposure within the context of psychological acceptance.
  Interventions: Behavioral: Exposure w/ Acceptance-Based Rationale
- Exposure w/ Habituation-Based Rationale (Active Comparator): Behavioral exposure within the context of habituation.
  Interventions: Behavioral: Exposure w/ Habituation-Based Rationale

INTERVENTIONS:
Behavioral: Exposure w/ Acceptance-Based Rationale — Treatment focuses on the ineffectiveness of participants' past attempts to control or reduce their anxiety in public speaking situations. Acceptance of one's private experiences (thoughts, feelings, sensations) will be introduced. "Willingness" to experience unwanted thoughts and feelings while simultaneously engaging in valued activities, especially those related to public speaking, is stressed. Techniques designed to foster psychological acceptance are practiced prior to and during exposure exercises, as well as assigned for homework between sessions.
  Arms: Exposure w/ Acceptance-Based Rationale
Behavioral: Exposure w/ Habituation-Based Rationale — Exposure to feared public speaking situations are accompanied by explanations of behavioral principles, including classical/operant conditioning and habituation. The process of associating public speaking situations with unwanted feelings of anxiety will be discussed, as well as negative reinforcement of escape and avoidance behaviors. The underlying principle of habituation is reviewed. When engaging in exposure exercises (both in session and assigned homework exercises), participants will be encouraged to remain in the feared speaking situation until their subjective ratings of anxiety decrease.
  Arms: Exposure w/ Habituation-Based Rationale

SUMMARY:
The purpose of this study is to compare two exposure-based behavioral group treatments for public speaking anxiety. Specifically, exposure within the context of psychological acceptance will be compared to exposure within a standard habituation context. It is hypothesized that participants receiving exposure within the context of psychological acceptance will experience a greater decrease in anxiety and greater improvement in quality of life compared to the habituation-based group.

DETAILED DESCRIPTION:
Social Anxiety Disorder (SAD) is a potentially debilitating condition affecting approximately 12% of the population at some point in their life (Ruscio et al., 2008). Nongeneralized SAD refers to individuals whose fears are limited to one or two social situations, most commonly public speaking. Empirically supported treatments for public speaking anxiety generally include an exposure component involving participation in anxiety-provoking public speaking situations (usually simulated situations using an audience of confederates and/or fellow participants, as well as actual public speaking situations in the community). Exposure is often presented within the context of habituation, but cognitively- based therapies utilize a rationale for exposure based on cognitive restructuring and belief modification. Research investigating the incremental benefit of adding other treatment components to exposure has yielded mixed results; however, there is preliminary evidence that the context in which exposure is presented can have an impact on treatment outcome. Recently, acceptance-based therapies have begun to frame exposure as an opportunity to increase one's willingness to experience anxiety while engaging in valued behaviors, rather than as a vehicle for modifying maladaptive cognitions and reducing anxiety. However, little research has been conducted on the efficacy of acceptance-based therapies for public speaking anxiety, and no component control studies have examined the utility of an acceptance/cognitive defusion rationale and context for exposure for public speaking anxiety. The present study will compare two exposure-based treatments for public speaking anxiety in a clinical sample. Specifically, exposure within an acceptance/defusion context will be compared to exposure with a habituation-based rationale.

Hypotheses:

1. Participants receiving exposure within an acceptance/defusion context will experience a greater reduction in anxiety and behavioral avoidance, and greater improvement in measures of quality of life, compared to participants receiving exposure within a habituation rationale, at post-treatment.
2. Acceptance, defusion, and mindfulness will mediate treatment outcome. Specifically, greater changes on measures of these three constructs will account for a significant portion of the effect of treatment condition on the dependent variables.
3. Lower baseline levels of public speaking anxiety and overall anxiety will be associated with higher baseline quality of life, mindfulness, acceptance, defusion, and social skills.
4. Baseline levels of acceptance, defusion, and mindfulness will predict overall treatment response, regardless of intervention condition.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosable public speaking anxiety (per DSM-IV-TR criteria for nongeneralized social anxiety disorder)
* Aged 18-65
* Residence in the greater Philadelphia area

Exclusion Criteria:

* Pervasive developmental disability
* Acute suicide potential
* Inability to travel to the treatment site
* Certain comorbid Axis I diagnoses, namely:

  * generalized SAD
  * schizophrenia or other psychotic disorder
  * current substance dependence
* Comorbid diagnoses of Major Depressive or other mood or anxiety disorders are acceptable ONLY if clearly secondary to the diagnosis of public speaking anxiety

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2009-02; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James D Herbert, Ph.D., Study Director — Drexel University; Evan M Forman, Ph.D., Study Director — Drexel University
Locations (1):
- Drexel University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] England, E.L., Herbert, J.D., Forman, E.M., Rabin, S.J., Juarascio, A., & Goldstein, S. (2012). Acceptance-based exposure therapy for public speaking anxiety. Journal of Contextual Behavioral Science, 1(1), 66-72.

RESULTS

PARTICIPANT FLOW:
Groups:
- Acceptance: Behavioral exposure within the context of psychological acceptance.
- Habituation: Behavioral exposure within the context of habituation.
Period: Overall Study
Arm/Group | Acceptance | Habituation
Started | 21 | 24
Completed | 16 | 19
Not Completed | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acceptance | Habituation | Total
Number analyzed (Participants) | 21 | 24 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 24 | 45
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.20 (12.40) | 29.96 (8.41) | 31.93 (10.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 36
  Male | 3 | 6 | 9
Region of Enrollment [Number; unit: participants]
  United States | 21 | 24 | 45

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in Remission (Per Structured Clinical Interview for DSM-IV Axis I Disorders (SCID))
Description: The SCID (First, Spitzer, Gibbon, & Williams, 1996) is an extensively utilized structured diagnostic interview based on DSM-IV criteria. Estimates of interrater reliability range from moderate to high for most Axis I disorders (e.g., Williams et al., 1992; Zanarini
  & Frankenburg, 2001).
Time Frame: 6-weeks post-treatment
Measure: Number; unit: participants
Arm/Group | Acceptance | Habituation
Number analyzed (Participants) | 21 | 24
participants | 21 | 20

ADVERSE EVENTS:
Arm/Group | Acceptance | Habituation
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/24
Other Adverse Events (participants affected / at risk) | 0/21 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No